CLINICAL TRIAL: NCT01068951
Title: Open Study to Evaluate the Safety and Efficacy of Autologous Mesenchymal Stem Cells in Treatment of Recently Diagnosed Patients With Type 1 Diabetes Mellitus
Brief Title: Treatment of Patients With Newly Onset of Type 1 Diabetes With Mesenchymal Stem Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Per-Ola Carlsson, Professor, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AS2010-0180
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; mesenchymal stem cells; intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- Mesenchymal stem cells (Active Comparator): Comparison of active treatment with autologous mesenchymal stem cells (in addition to standard treatment) to standard treatment of patients newly diagnosed with type 1 diabetes mellitus.
  Interventions: Biological: Mesenchymal stem cells
- Control (No Intervention)

INTERVENTIONS:
Biological: Mesenchymal stem cells — Autologous transplantation of the patients own mesenchymal stem cells (approximately 2 x 106 cells/kg body weight) intravenously.
  Arms: Mesenchymal stem cells

SUMMARY:
The main hypothesis of the investigators study is that the development of autoimmune diabetes may be halted att diagnosis by the immune modulatory properties of mesenchymal stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Mentally stable and able to comply with the procedures of the study protocol
* Clinical history compatible with type 1 diabetes diagnosed less than 10 days of enrolment Stimulate c-peptide >0.1 nmol/l

Exclusion Criteria:

* Patients with BMI>30
* Patients with unstable cardiovascular status
* Patients with active infections, unless treatment is not judged necessary by the investigators
* Patients with serological evidence of infection with HIV, hepatitis B or hepatitis C.
* Sexually active females who are not a) postmenopausal, b) surgically sterile or c) using an acceptable method of contraception: oral contraceptives, Norplant, Depo-provera and barrier devices combined with spermicidal gel are acceptable.
* Patients with known or previous malignancy. Patient with any condition or any circumstance that in the opinion of the investigator would make it unsafe to undergo treatment with autologous MSC.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The concentration of stimulated c-peptide at 90 minutes after the start of a mixed meal tolerance test at 365+/-10 days following the infusion or not with mesenchymal stem cells | 1 year after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Carlsson PO, Schwarcz E, Korsgren O, Le Blanc K. Preserved beta-cell function in type 1 diabetes by mesenchymal stromal cells. Diabetes. 2015 Feb;64(2):587-92. doi: 10.2337/db14-0656. Epub 2014 Sep 9. PMID 25204974